CLINICAL TRIAL: NCT06845813
Title: A Phase I, Multicentre, Single-Dose, Non-Randomised, Open-Label, Parallel-Group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD6234
Brief Title: Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD6234
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8750C00007
Record Dates: First submitted 2025-02-24; First posted 2025-02-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Healthy Participants; AZD6234; Pharmacokinetics; Safety
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Up to five cohorts (four renal impairment cohorts and controls with normal renal function) will be enrolled into the study.
  All subjects will receive the study intervention:
  * Cohort 1 will enroll participants with end stage renal disease
  * Cohort 2 will enroll participants with severe renal impairment
  * Cohort 3 will enroll healthy participants matched on a group level by sex, age, and BMI
  * Cohort 4 (optional) will enroll participants with moderate renal impairment
  * Cohort 5 (optional) will enroll participants with mild renal impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Subjects with end stage renal disease will receive a single subcutaneous dose of AZD6234 under fasted conditions
  Interventions: Drug: AZD6234
- Group 2 (Experimental): Subjects with severe renal impairment will receive a single subcutaneous dose of AZD6234 under fasted conditions
  Interventions: Drug: AZD6234
- Group 3 (Experimental): Healthy participants will receive a single subcutaneous dose of AZD6234 under fasted conditions
  Interventions: Drug: AZD6234
- Group 4 (optional) (Experimental): Subjects with moderate renal impairment will receive a single subcutaneous dose of AZD6234 under fasted conditions
  Interventions: Drug: AZD6234
- Group 5 (optional) (Experimental): Subjects with mild renal impairment will receive a single subcutaneous dose of AZD6234 under fasted conditions
  Interventions: Drug: AZD6234

INTERVENTIONS:
Drug: AZD6234 — Dose 1
  Other Names: Dose 1

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of single subcutaneous dose of AZD6234 with end stage renal disease, severe, and possibly moderate and mild renal impairment in comparison to a matched healthy control group.

DETAILED DESCRIPTION:
This Phase I multicentre, single-dose, non-randomised, open-label, parallel-group study aims to examine the pharmacokinetics, safety, and tolerability of AZD6234 in both male and female participants. Participants include those with end-stage renal disease (ESRD) on intermittent haemodialysis (HD), severe renal impairment not on dialysis, and optional groups for moderate and mild renal impairment. These are compared to participants with normal renal function. All participants are grouped based on body surface area-adjusted estimated glomerular filtration rate (eGFR), and those with normal renal function are matched at a group level by sex, age, and body mass index (BMI) to the participants with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 85 years of age, inclusive, at the time of signing the informed consent.
* Body weight ≥ 50 kg; BMI within the range of ≥ 18 to ≤ 40 kg/m2, as measured at screening.

Healthy Matched Control Participants:

* Participant must be medically healthy with no clinically significant medical history, or abnormalities in physical examination, clinical laboratory profiles, vital signs, or 12-lead ECGs, as deemed by the investigator at screening and Day -1.
* Have an eGFR of ≥ 90 mL/min determined at screening.

Renally-impaired Participants:

* Diagnosis of chronic kidney disease, stable renal function in the 3 months prior to dosing,
* Participants with renal impairment based on BSA-adjusted CKD-EPI equation at screening.
* All renally-impaired participants should be on a stable dose of cardio-renal relevant treatment for at least 2 weeks prior to screening.
* If participants with renal impairment have diabetes mellitus, it must be controlled
* Female(s) of childbearing potential: must use adequate contraception. Oral contraceptives are not permitted as there is a potential effect of the IMP on the absorption of oral drugs.
* Male Participants: Condom use is required for the duration of the study and until at least 28 days after the last dose of IMP. Additional contraception must be used for the sexual partners of male study participants throughout the clinical trial and for 28 days following the last dose of IMP.

Exclusion Criteria:

- History or presence of: significant GI disease or previous upper GI surgery

* Clinically significant cardiovascular disease, as judged by the investigator, d. Neuromuscular or neurogenic disease e. Severe vitamin D deficiency < 12 ng/dL.
* History or presence of any condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of psychosis, bipolar disorder
* History of major depressive disorder within the past 2 years
* History of suicide attempt or history of suicidal ideation within the past year.

Healthy Matched Control Participants:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* Use of any prescription or non-prescription drugs, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.

Renally-impaired Participants:

* Presence of unstable medical condition or any evidence of additional severe or uncontrolled systemic disease or laboratory finding which, in the opinion of the investigator, would compromise the participant's safety or successful participation in this study.
* Renal transplant patients, participants waiting for organ transplant scheduled to occur during the study, and those with a history of acute kidney injury occurring within 3 months prior to screening. Nonfunctioning renal allografts are allowed.
* Use of concurrent medication which affects calculation of eGFR by affecting serum creatinine within 7 days of Day -1.
* Unable to refrain from phosphate binders, cholestyramine/colestipol, and ranitidine/nizatidine within 10 hours before and 10 hours after study intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
AUClast | Day 1 to Day 36
  Area under plasma concentration-time curve from time zero to the last measurable concentration
AUCinf | Day 1 to Day 36
  Area under plasma concentration-time curve from zero to infinity
Cmax | Day 1 to Day 36
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 36
  Time to reach maximum observed plasma concentration
PK parameter (t1/2λz) | Day 1 to Day 36
  Terminal elimination half-life
PK parameter (CL/F) | Day 1 to Day 36
  Apparent plasma clearance
PK parameter (Vz/F) | Day 1 to Day 36
  Apparent volume of distribution during the terminal phase
Number of participants with adverse events (AEs) | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.
Number of participants with abnormal vital signs | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.
Number of participants with abnormal ECGs | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.
Number of participants with abnormal physical examination findings | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.
Number of participants with abnormal laboratory test results | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.
Number of participants with confirmed positive anti-drug antibody testing | Day 1 to Day 54
  Prevalence and incidence of ADAs to AZD6234 ADA titre
Number of participants with serious adverse events (SAEs) | Day 1 to Day 54
  To assess the safety and tolerability of a single subcutaneous dose of AZD6234 in participants with end stage renal disease, severe, moderate (optional), and mild (optional) renal impairment and those with normal renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Saba, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares; Thomas C Marbury, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares; Joel M Neutel, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares; Kwabena Ayesu, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares
Locations (2):
- United States (2):
  - Research Site, Lake Forest, California
  - Research Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home